CLINICAL TRIAL: NCT04603157
Title: Remote Self-training Program for Patients With Postural Orthostatic Tachycardia Syndrome (POTS)
Brief Title: Remote Self-training Program for Patients With Postural Orthostatic Tachycardia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Courtney M. Wheatley, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-007186
Record Dates: First submitted 2020-10-15; First posted 2020-10-26 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Group (No Intervention): Subject with diagnosed with postural orthostatic tachycardia syndrome will continue to follow the treatment recommendations of the primary care physician
- Hybrid Exercise Training Group (Experimental): Subject with diagnosed with postural orthostatic tachycardia syndrome will follow a hybrid exercise training program
  Interventions: Behavioral: Hybrid Exercise Training

INTERVENTIONS:
Behavioral: Hybrid Exercise Training — Personalized exercise program completing at least 3 aerobic exercise sessions a week and receive eight supervised training sessions over the 3-months
  Arms: Hybrid Exercise Training Group

SUMMARY:
The purpose of this research is to evaluate if a hybrid semi-supervised remote exercise training program can reduce symptoms and improve quality of life and physical fitness in individuals with postural orthostatic tachycardia syndrome (POTS) and determine if this program is more effective than current standard of care.

DETAILED DESCRIPTION:
To answer these questions, 60 individuals with POTS will be recruited to complete a symptom-limited cardiopulmonary exercise test with measures of cardiac output, autonomic function testing, blood volume measurement, and QOL questionnaires at baseline and following 3-months of treatment. Thirty participants will be randomized to continue with the standard of care which can include lower body and core strengthening, fluids, salt, medications and sometimes exercise. The other thirty participants will be asked to complete at least three exercise training sessions a week (progressing to 3hrs/wk of aerobic and 1hr/wk of strength training) and receive eight supervised training sessions over the 3-month treatment period. All participants will be provided with a polar heart rate monitor which will be linked to a connected health application to allow patients to track any aerobic workout, ensure during a session they are in the correct training zone, and allow the study team to remotely monitor adherence.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years old or older
* Meet diagnosis criteria for POTS = a heart rate increase of ≥ 30bpm with supine to 10 minutes of standing or head-up tilt or heart rate exceeding 120 ppm after 10 minutes of standing or tilt without evidence of orthostatic hypertension (a fall in BP of > 20/10 mmHg)
* Been diagnosed with POTS ≥6 months prior to participation in the study (chronic)
* Female subjects must not be pregnant or trying to become pregnant during duration of study participation
* Those in exercise training group must be on stable medications for at least 1 month and medication must remain consistent for duration of study participation. For those in the standard of care group, a change in medication will be allowed within the first month following baseline testing, but then must remain consistent until 3-month testing time point.
* Ehlers-Danlos Syndrome (EDS) patients will be included, but will target equal randomization between treatment groups

Exclusion Criteria:

* Individual is not eligible if they are currently exercising, cut off >30 minutes of structured exercise/physical activity per week. (assessed by Global Physical Activity Questionnaire)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Change Peak Oxygen consumption at 3 months | baseline and following 3 month intervention
  peak oxygen consumption measured from maximal cardiopulmonary exercise testing

SECONDARY OUTCOMES:
Change in Composite Autonomic Symptom Score (COMPASS 31) at 3 months | baseline and following 3 month intervention
  Composite Autonomic Symptom Score a questionnaire of autonomic symptoms severity in 6 domains. Total score ranges from 0-100. Higher score means more severe autonomic symptoms.
Change in Functional Ability Score at 3 months | baseline and following 3 month intervention
  Functional Ability Score asking patient to report their degree of limitation from 0-100% in 10% increments. 100% would be no limitation, feel normal, 10% is completely bedridden.
Change in 36-Item Short Form Health Survey questionnaire (SF-36) at 3 months | baseline and following 3 month intervention
  36-Item Short Form Health Survey questionnaire to evaluate quality of life and degree of health specifically focusing on the reported physical and mental components. Scores range from 0-100, where a higher score indicated better health.
Change in heart rate with 10-min Stand test at 3 months | baseline and following 3 month intervention
  Change in heart rate in response to standing from supine to standing for 10 minutes
Change in blood volume at 3 months | baseline and following 3 month intervention
  change in blood volume

OTHER OUTCOMES:
Change in anaerobic threshold oxygen consumption at 3 months | baseline and following 3 month intervention
  Change in oxygen consumption at anaerobic threshold measured from maximal cardiopulmonary exercise testing
Change in matched workload oxygen consumption at 3 months | baseline and following 3 month intervention
  Change in oxygen consumption at matched workload measured from maximal cardiopulmonary exercise testing
Change in anaerobic threshold heart rate at 3 months | baseline and following 3 month intervention
  Change in heart rate at anaerobic threshold measured from maximal cardiopulmonary exercise testing
Change in matched workload heart rate at 3 months | baseline and following 3 month intervention
  Change in heart rate at matched workload measured from maximal cardiopulmonary exercise testing
Change in anaerobic threshold workload at 3 months | baseline and following 3 month intervention
  change in workload at anaerobic threshold measured from maximal cardiopulmonary exercise testing
Change in anaerobic threshold rating of perceived exertion (RPE) at 3 months | baseline and following 3 month intervention
  change in RPE at anaerobic threshold measured from maximal cardiopulmonary exercise testing
Change in matched workload rating of perceived exertion (RPE) at 3 months | baseline and following 3 month intervention
  Change in RPE at matched workload measured from maximal cardiopulmonary exercise testing
Change in anaerobic threshold cardiac output at 3 months | baseline and following 3 month intervention
  change in cardiac output at anaerobic threshold measured from maximal cardiopulmonary exercise testing
Change in matched workload cardiac output at 3 months | baseline and following 3 month intervention
  Change in cardiac output at matched workload measured from maximal cardiopulmonary exercise testing

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Wheatley-Guy, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials